CLINICAL TRIAL: NCT07243431
Title: Pediatric Medication Safety Revolution: Auditing Nurses' Knowledge on High-Alert Drugs
Brief Title: Knowledge About the Administration and Regulation of High Alert Medications Among Nurses in Mansoura University Children's Hospital: A Hospital-wide Audit
Acronym: HAM-Audit
Status: Completed | Type: Observational
Sponsor: Omar Hamdy (Other)
Responsible Party: Sponsor-Investigator, Omar Hamdy, prof, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: R.25.01.3028
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Nurses' Knowledge of High-alert Medications in Pediatric Care
Keywords: high-alert medications; nurses knowledge; medication errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study checks how well nurses at Mansoura University Children's Hospital know about high-alert medications (HAMs). These are drugs that can cause serious harm if given incorrectly. We used a questionnaire to assess their knowledge and identify any gaps. The goal is to improve training and reduce medication errors in the hospital.

DETAILED DESCRIPTION:
Background:

Medication errors (MEs) are a major cause of patient harm, especially in pediatric settings. High-alert medications (HAMs) are drugs that carry a heightened risk of causing significant patient harm when used in error. Nurses play a critical role in the safe administration of HAMs. This hospital-wide audit aims to evaluate nurses' knowledge regarding the administration and regulation of HAMs at Mansoura University Children's Hospital.

Objectives:

1. To assess the level of knowledge about HAMs among nurses.
2. To identify factors associated with sufficient knowledge of HAMs.

Methods:

A cross-sectional study was conducted using a self-administered questionnaire distributed to all nurses involved in medication administration at Mansoura University Children's Hospital. The questionnaire covered identification of HAMs, storage, administration protocols, and error prevention strategies. Data was collected from [February to October 2025] and analyzed using descriptive statistics and logistic regression.

Setting:

Mansoura University Children's Hospital, Mansoura, Egypt.

Participants:

All registered nurses working in the hospital and involved in medication administration.

Outcome Measures:

* Primary: Level of knowledge about HAMs (scored as sufficient/insufficient).
* Secondary: Factors associated with sufficient knowledge (e.g., years of experience, training).

ELIGIBILITY:
Inclusion Criteria:

* - Registered nurses working at Mansoura University Children's Hospital.
* Involved in medication administration.
* At least 6 months of experience in the hospital.

Exclusion Criteria:

* Non-nursing staff.
* Nurses not involved in direct patient care or medication administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All registered nurses working at Mansoura University Children's Hospital who are involved in medication administration. The study includes nurses from various departments with at least 6 months of experience. This hospital-wide audit targets frontline healthcare providers responsible for high-alert medication handling in a tertiary pediatric setting.
Sampling Method: Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Proportion of nurses with sufficient knowledge of high-alert medications | February 2025 to October 2025
  Percentage of nurses scoring ≥70% on the questionnaire assessing knowledge of high-alert medications (identification, administration, storage, and error prevention).

SECONDARY OUTCOMES:
Factors associated with sufficient knowledge of high-alert medications | February 2025 to October 2025
  Identification of factors (e.g., years of experience, training, department) associated with scoring ≥70% on the knowledge questionnaire using multivariate logistic regression.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children's Hospital, Al Mansurah, Egypt